CLINICAL TRIAL: NCT01606085
Title: Cost Effectiveness and Quality of Life in Heart Failure Patients With Diabetes
Acronym: QUALITYHF-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency); Atlanta Clinical and Translational Science Institute (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sandra B. Dunbar, RN, Professor and Associate Dean of Academic Advancement, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00026671; 1R01NR011888-01 (NIH)
Record Dates: First submitted 2012-05-14; First posted 2012-05-25 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus; Heart Failure
Keywords: Diabetes; Heart Failure; Quality of Life; Self Care
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HF-DM Self Care (Experimental): educational counseling intervention about integrated HF-DM self care outcomes
  Interventions: Behavioral: HF DM self care; Behavioral: Usual Care
- Usual Care (No Intervention): Usual Care provided by providers

INTERVENTIONS:
Behavioral: HF DM self care — Education in monitoring signs and symptoms of Heart Failure and Diabetes as well as self care instruction
  Other Names: HF-DM Self Care
  Arms: HF-DM Self Care
Behavioral: Usual Care — Educational materials on Heart Failure and diabetes at study enrollment. Full educational binder delivered at end of study.
  Arms: HF-DM Self Care

SUMMARY:
The purposes of this study are:

1. to develop and test an integrated self care intervention for Heart Failure (HF)patients with Diabetes (DM) for its effects on patient outcomes including health related quality of life (HRQOL), physical function and health resource utilization.
2. to assess the costs and cost effectiveness of the intervention.

The intervention is designed to go beyond usual care of providing separate Heart Failure (HF) and Diabetes (DM) patient education by educating HF-DM patients on integrated self care and self management related to a HF-DM diet, HF-DM medication-taking behaviors, physical activity, and HF-DM symptom monitoring and management. An integrated self care intervention will compare HF-DM patients who receive the intervention with those who receive usual care-attention control for effects on patient outcomes,self care process measures, and health care utilization. If effective, the intervention will lead to improved self care, improved quality of life, and reduced health care resource use and costs. This study will facilitate greater understanding of self care within the context of two chronic illnesses and will lead directly to improved clinical practice and future research on comorbid self care in Heart Failure.

DETAILED DESCRIPTION:
The investigators hypothesize that participants receiving the Heart Failure and Diabetes (HF-DM) self-care intervention will report greater Health Related Quality of Life (HRQOL) on the Minnesota Living with HF Questionnaire (MLHFQ), the Audit of Diabetes-dependent Quality of Life (ADDQoL), and the EuroQol (EQ5D) than the Usual Care (UC-AC) group at 6 months when controlling for age, gender, and NYHA Class.

Secondly, that participants receiving the Heart Failure and Diabetes (HF-DM) self-care intervention will demonstrate improved physical function indicators (BNP levels, HgA1c, and 6MWT) at 6 months over the UC-AC group when controlling for age, gender, BMI, and NYHA Class and comorbid conditions.

Thirdly, that participants receiving the Heart Failure and Diabetes (HF-DM) self-care intervention will exhibit greater improvement in: HF knowledge and DM knowledge than UC-AC at 6 months. Participants receiving the integrated HF-DM self-care intervention will report greater improvements in HF self-efficacy and DM self-efficacy over UC-AC at 6 months. HF-DM patients randomized to the integrated self-care intervention will exhibit greater improvements in overall HF and DM self-care behaviors and HF-DM diet and physical activity over UC-AC at 6 months.

Lastly, that HF-DM patients who receive the integrated self-care intervention will exhibit less health resource use and associated costs(direct health care costs of provider visits, hospitalizations, ED visits, length of stay, and direct non-health care costs associated with the HRU and intervention) over the 6 months than those who receive UC-AC controlling for comorbidity and insurance status.

ELIGIBILITY:
Inclusion Criteria:

* hospital admission with a diagnosis of Heart Failure (HF) with Left Ventricular Systolic Dysfunction (LVSD) or diastolic dysfunction and concomitant Diabetes (DM) type II
* planned discharge from hospital to home setting
* NYHA Class II-IV
* On optimal HF regimen of care including ACE-Inhibitors or ARBs beta blocking agents, and diuretics if indicated by patient fluid status
* ambulatory
* able to read and write English
* acceptable cognitive screening test

Exclusion Criteria:

* planned discharge to long term acute care
* presence of an insulin pump
* active foot ulcer
* presence of hemodynamically significant angina pectoris
* renal failure with hemodialysis
* planned cardiac surgery
* impaired cognition due to neurological comorbidity
* psychiatric diagnosis
* uncorrected visual or hearing problem
* uncorrected hearing or vision problems
* moderately severe depressive symptoms
* UNOS/ A status or ventricular assist device
* lack of telephone access

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Heart failure health related quality of life measures | 6 months
  As measured by Minnesota Living with Heart Failure Questionnaire (MLHFQ).
Diabetes health related quality of life measures | 6 months
  As measured by Audit of Diabetes - Dependent Quality of Life (ADDQOL).

SECONDARY OUTCOMES:
Heart Failure and Diabetes (HF-DM) physical outcomes | 6 months
  BNP and HgA1c, and 6 minute walk test
Heart Failure Knowledge | 6 months
  As measured by the Atlanta Heart Failure Knowledge Test (AHFKT)
Health resource use | 6 months
  As measured by hospital and ED visits as well as contact with medical providers
Heart Failure (HF) self-efficacy | 6 months
  As measured by Self Care in Heart Failure Inventory Self Efficacy Scale
Heart Failure and Diabetes(HF-DM) self-care behaviors | 6 months
  As measured by activity calendars/logs, Self care in Heart failure Inventory subscales, and Summary of Diabetes Self Care Scale
Diabetes (DM) Knowledge | 6 months
  Michigan Diabetes Knowledge Test (MDKT)
Diabetes (DM) self efficacy | 6 months
  Measured by the Perceived Diabetes Self Management Scale (PDSMS)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Dunbar, PhD, Principal Investigator — Nell Hodgson Woodruff School of Nursing; Javed Butler, MD, Study Director — Emory University; Stephen Culler, MD, Study Director — Emory University; Rebecca A. Gary, PhD, Study Director — Nell Hodgson Woodruff School of Nursing; Carolyn M. Reilly, PhD, Study Director — Nell Hodgson Woodruff School of Nursing
Locations (1):
- Emory University School of Nursing, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Reilly CM, Butler J, Culler SD, Gary RA, Higgins M, Schindler P, Butts B, Dunbar SB. An economic evaluation of a self-care intervention in persons with heart failure and diabetes. J Card Fail. 2015 Sep;21(9):730-7. doi: 10.1016/j.cardfail.2015.06.382. Epub 2015 Jul 8. PMID 26164214
- [Derived] Dunbar SB, Reilly CM, Gary R, Higgins MK, Culler S, Butts B, Butler J. Randomized clinical trial of an integrated self-care intervention for persons with heart failure and diabetes: quality of life and physical functioning outcomes. J Card Fail. 2015 Sep;21(9):719-29. doi: 10.1016/j.cardfail.2015.05.012. Epub 2015 May 29. PMID 26028261